CLINICAL TRIAL: NCT06062420
Title: A Phase 2, Randomized, Open-label, Platform Study Using a Master Protocol to Evaluate Novel Immunotherapy Combinations as First-Line Treatment in Participants With Recurrent/Metastatic PD-L1 Positive Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Platform Study of Novel Immunotherapy Combinations as First-Line Treatment in Participants With PD-L1 Positive Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck- GALAXIES H&N-202
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: iTeos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219885; 2023-503428-24 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-09-21; First posted 2023-10-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms, Head and Neck
Keywords: Dostarlimab; Belrestotug; Nelistotug; Remzistotug; PD-L1; HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dostarlimab Monotherapy (Experimental)
  Interventions: Drug: Dostarlimab
- Sub study 1: Dostarlimab and Belrestotug (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Belrestotug
- Sub study 2: Dostarlimab and nelistotug (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Nelistotug
- Sub study 3: Dosarlimab and Belrestotug and nelistotug (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Belrestotug; Drug: Nelistotug
- Sub study 4: Dostarlimab and remzistotug (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Remzistotug

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab will be administered.
Drug: Belrestotug — Belrestotug will be administered.
  Arms: Sub study 1: Dostarlimab and Belrestotug; Sub study 3: Dosarlimab and Belrestotug and nelistotug
Drug: Nelistotug — Nelistotug will be administered.
  Arms: Sub study 2: Dostarlimab and nelistotug; Sub study 3: Dosarlimab and Belrestotug and nelistotug
Drug: Remzistotug — Remzistotug will be administered.
  Arms: Sub study 4: Dostarlimab and remzistotug

SUMMARY:
The primary purpose of the study is to evaluate the antitumor activity and safety of novel immunotherapy combinations compared with dostarlimab in participants with Programmed death ligand 1 (PD-L1) positive Recurrent/Metastatic (R/M) Head and Neck Squamous Cell Carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically-confirmed HNSCC that is R/M and is considered incurable by local therapies. A) Subjects must not have had prior systemic therapy administered in the R/M setting. Chemoradiation therapy which was completed more than 4 months prior to signing consent if given as part of multimodal treatment for locally advanced disease is allowed B) The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx C) Subjects may not have a primary tumor site of nasopharynx (any histology)
* Has measurable (target) disease based on RECIST 1.1 as determined by the investigator.
* Has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Provides a tumor tissue sample obtained at the time of or after the initial diagnosis of R/M HNSCC. A fresh tumor tissue sample obtained within 90 days of screening is highly preferred, If fresh biopsy is not possible, an archival tumor specimen is acceptable unless it was obtained prior to administration of chemoradiation for the treatment of a participant's tumor. Needle or excisional biopsies or resected tissue is required. Cytological specimens such as fine needle aspirates, bone marrow samples, or cell blocks are not acceptable. Bone specimen is not acceptable.
* Has tumor Programmed death ligand 1 (PD-L1) expression
* If the primary tumor site is oropharyngeal carcinoma, the participant must have Human papillomavirus (HPV) results

Exclusion Criteria:

* Has received prior therapy with any immune checkpoint inhibitors, including antibodies or drugs targeting Programmed death protein 1 (PD-1), PD-L1, Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), T cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine based inhibitory motif domains (TIGIT), Cluster of differentiation (CD) 96, or other immune checkpoint pathways.
* Participants with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, esophageal, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
* Have active tumor bleeding or a high risk of bleeding (examples include but are not limited to radiographic evidence of major blood vessel invasion/infiltration or tumor demonstrates >90 degree abutment or encasement of a major vessel [carotid, jugular, bronchial artery] and/or exhibits other high-risk features such as arteriovenous fistula).
* Has PD within 4 months of completion of curatively intended treatment for locoregionally advanced HNSCC
* Participants with any carcinomatous meningitis or leptomeningeal spread and those with uncontrolled or symptomatic Central Nervous System (CNS) metastases
* Active autoimmune disease that has required systemic disease-modifying or immunosuppressive treatment within the last 2 years. (Stable, medically managed autoimmune endocrinopathies are acceptable if participant otherwise meets entry criteria.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) compared between Sub studies and Dostarlimab monotherapy | Up to approximately 24 months
  Confirmed ORR is defined as the percentage of participants achieving confirmed Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator assessment.

SECONDARY OUTCOMES:
Rate of Circulating Tumor Deoxyribonucleic Acid (ctDNA) Molecular Response | Up to approximately 24 months
  The rate of ctDNA molecular response, is defined as the percentage of participants achieving a ≥50% decrease in ctDNA level compared to baseline, measured by plasma ctDNA assessment.
Number of Participants with Treatment Emergent Adverse Events (AEs), treatment emergent Serious Adverse Events (SAE) and treatment emergent Adverse Events of Special Interest (AESI) | Up to approximately 24 months
Number of Participants with TEAEs leading to dose modifications or study intervention discontinuation | Up to approximately 24 months
Number of Participants with Clinically Significant Findings in Vital signs, Electrocardiogram (ECG), and Laboratory test parameters | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (96):
- United States (5):
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (8):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Florida
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, Santa Fe
- Brazil (2):
  - GSK Investigational Site, Santo André
  - GSK Investigational Site, São Paulo
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Herlev, Denmark
- GSK Investigational Site, Turku, Finland
- France (6):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Villejuif
- Germany (9):
  - GSK Investigational Site, Aachen
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Giessen
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Regensburg
  - GSK Investigational Site, Ulm
- Greece (3):
  - GSK Investigational Site, Haidari - Athens
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kecskemét
  - GSK Investigational Site, Pécs
- Italy (10):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Novara
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
- Japan (7):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Oslo, Norway
- Poland (7):
  - GSK Investigational Site, Bielsko-Biala
  - GSK Investigational Site, Gliwice
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Przemyśl
  - GSK Investigational Site, Siedlce
  - GSK Investigational Site, Warsaw
- Portugal (3):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Romania (8):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Suceava
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do
- Spain (8):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Taiwan (3):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/